CLINICAL TRIAL: NCT05516316
Title: A Randomised, Double-blind, Placebo-controlled Proof-of-pharmacology Study of EP395 in Healthy Adults
Brief Title: Clinical Trial Comparing the Pharmacological Effects of EP395 With Placebo in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EpiEndo Pharmaceuticals (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EP395-002; 2021-005867-28 (EudraCT Number)
Record Dates: First submitted 2022-08-16; First posted 2022-08-25 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: The study is double-blind, placebo-controlled and parallel-group in design.
Who Masked: Participant, Investigator
Masking Description: During the study, study participants, investigators, the sponsor, and all other persons involved in the conduct of the study will be blinded to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EP395 high dose (Experimental): EP395 in repeated doses. Orally, once-daily administration of 3 EP395 capsules for 21 days
  Interventions: Drug: EP395
- EP395 low dose (Experimental): EP395 in repeated doses. Orally, once-daily administration of 1 EP395 capsule and 2 placebo capsules for 21 days
  Interventions: Drug: EP395
- Placebo (Placebo Comparator): Matched placebo capsule, once-daily administration of 3 placebo capsules for 21 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EP395 — Capsule for oral use
  Arms: EP395 high dose; EP395 low dose
Drug: Placebo — Capsule for oral use
  Arms: Placebo

SUMMARY:
This study aims to assess the effect of EP395 against an induced inflammation of the lung. In addition, further data about the safety and tolerability of EP395 will be collected.

To investigate the efficacy of EP395 at the end of the treatment with EP395 or placebo (dummy), all participants will inhale a lipopolysaccharide (a molecule composed of sugar and fat) that artificially induces an acute inflammation of the airways. It is assumed that participants who received EP395 will show less inflammation of the airways than participants who received placebo.

DETAILED DESCRIPTION:
This is a study to assess the pharmacological effect of repeated doses of EP395 in healthy subjects with the aim to assess the effects of EP395 on lung and blood markers of inflammation after inhaled lipopolysaccharide (LPS), and the safety, tolerability, and systemic exposure of EP395.

The study will be randomised in a 1:1 ratio to take either high dose EP395 or placebo as oral capsules once daily for 21 days starting on Day 1 with scheduled visits at Days 7, 14, and 21 for assessments of safety and tolerability and systemic exposure of EP395. At Day 21, 2 hours after the last investigational product (IP) intake, participants will undergo an inhaled LPS challenge to induce airway inflammation, which will be followed by bronchoscopy and BAL 6 hours later. A final safety follow-up visit will be performed at Day 37.

If the data from the high dose EP395 arm (variability, effect size) indicate that it may be possible to detect effects on IL-8 at a lower dose of EP395, an additional lower dose EP395 arm will be added.

ELIGIBILITY:
1. Willing and able to understand the information on the nature, the scope and the relevance of the clinical study, and to provide voluntary, written informed consent to participate in the study before any study-related procedures
2. Men and women, aged ≥18 and ≤55 years
3. Women of childbearing potential must:

   1. have a negative pregnancy test (blood) at Screening.
   2. agree to use, and be able to comply with, highly effective measures of contraceptive control (failure rate less than 1% per year when used consistently and correctly) without interruption, from Screening until 90 days after the last IP intake.
4. Men must agree to use contraception (barrier method) during sexual intercourse with women of childbearing potential during treatment until 90 days after the last IP intake and should not donate sperm during this time.
5. In good health as determined by medical history and screening investigations, as judged by the investigator
6. Body mass index of ≥19 and ≤33 kg/m2
7. Normal spirometry (forced expiratory volume in 1 second [FEV1] >80% predicted and FEV1/forced vital capacity >70%)
8. Non-smoker or former smoker with <10 pack years who had stopped smoking (including e-cigarettes) for at least 6 months before Screening.

Exclusion Criteria:

1. History or presence of any clinically relevant medical condition that could affect the participant's safety or interfere with the objectives of the study
2. Presence or history of lung disease, eg, asthma, chronic obstructive pulmonary disease
3. Clinically significant abnormality on 12-lead ECG including prolonged corrected QT interval by Fredericia (>450 msec men or >470 msec women)
4. Use of prescribed or nonprescribed medications or herbal remedies within 28 days of first dosing and during the study with the exception of

   1. hormone replacement therapy (HRT)
   2. contraception
   3. occasional use of paracetamol
5. Positive hepatitis B surface antigen, hepatitis C antibodies, HIV-1 or -2 antibodies
6. Positive drugs of abuse, smoking, or alcohol test at Screening
7. History of alcohol or drug misuse
8. Pregnant and lactating women
9. Prior recovery from recent infection, including but not limited to COVID-19, within the last 14 days before first dosing with IP
10. History of hypersensitivity to any constituents of the IMP or LPS
11. Any clinically significant allergy
12. Participation in a clinical study with an IP within 3 months or 5 half-lives before first dosing, whichever is longer
13. Employees of the sponsor or employees or relatives of the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Bronchoalveolar lavage fluid interleukin 8 at Day 21 | Day 21

SECONDARY OUTCOMES:
ECG ventricular rate | Screening (Day -21 to Day -1), Days 1, 7 (±2 days), 14 (±2 days), Day 21 (±2 days), Day 37 (±3 days)
  Absolute values and changes from baseline will be summarized for all assessed time points
ECG RR interval | Screening (Day -21 to Day -1), Days 1, 7 (±2 days), 14 (±2 days), Day 21 (±2 days), Day 37 (±3 days)
  Absolute values and changes from baseline will be summarized for all assessed time points
ECG PR interval | Screening (Day -21 to Day -1), Days 1, 7 (±2 days), 14 (±2 days), Day 21 (±2 days), Day 37 (±3 days)
  Absolute values and changes from baseline will be summarized for all assessed time points
ECG QRS duration | Screening (Day -21 to Day -1), Days 1, 7 (±2 days), 14 (±2 days), Day 21 (±2 days), Day 37 (±3 days)
  Absolute values and changes from baseline will be summarized for all assessed time points
ECG QT interval (uncorrected) | Screening (Day -21 to Day -1), Days 1, 7 (±2 days), 14 (±2 days), Day 21 (±2 days), Day 37 (±3 days)
  Absolute values and changes from baseline will be summarized for all assessed time points
ECG QTcF intervals | Screening (Day -21 to Day -1), Days 1, 7 (±2 days), 14 (±2 days), Day 21 (±2 days), Day 37 (±3 days)
  Absolute values and changes from baseline will be summarized for all assessed time points
Assessment of laboratory values (haematology) | Screening (Day -21 to Day -1), Days 1, 7 (±2 days), 14 (±2 days), Day 21 (±2 days), Day 37 (±3 days)
  Absolute values and changes from baseline will be summarized for all assessed time points
Assessment of laboratory values (blood biochemistry) | Screening (Day -21 to Day -1), Days 1, 7 (±2 days), 14 (±2 days), Day 21 (±2 days), Day 37 (±3 days)
  Absolute values and changes from baseline will be summarized for all assessed time points
Assessment of blood coagulation | Screening (Day -21 to Day -1), Days 1, 7 (±2 days), 14 (±2 days), Day 21 (±2 days), Day 37 (±3 days)
  Absolute values and changes from baseline will be summarized for all assessed time points
Urinalysis | Screening (Day -21 to Day -1), Days 1, 7 (±2 days), 14 (±2 days), Day 21 (±2 days), Day 37 (±3 days)
  Absolute values and changes from baseline will be summarized for all assessed time points
Vital signs: Systolic and diastolic blood pressure | Screening (Day -21 to Day -1), Days 1, 7 (±2 days), 14 (±2 days), Day 21 (±2 days)
  Absolute values and changes from baseline will be summarized for all assessed time points
Vital signs: Pulse | Screening (Day -21 to Day -1), Days 1, 7 (±2 days), 14 (±2 days), Day 21 (±2 days)
  Absolute values and changes from baseline will be summarized for all assessed time points
Vital signs: Body temperature | Screening (Day -21 to Day -1), Days 1, 7 (±2 days), 14 (±2 days), Day 21 (±2 days)
  Absolute values and changes from baseline will be summarized for all assessed time points
Height and weight | Screening (Day -21 to Day -1), Day 37 (±3 days)
  BMI will be calculated from height and weight measurements
Standard routine physical examination | Screening (Day -21 to Day -1), Days 1, Day 21 (±2 days), Day 37 (±3 days)
  A standard routine physical body examination will be performed and abnormal physical examination results will be evaluated and reported as AEs.
Assessment of adverse event (AE) occurrence | From Screening (Day -21 to Day -1), to Day 37 (±3 days)
BALF cell count (total and differential) and mediators | Day 21 (±2 days)
  Including tumour necrosis factor (TNF)-α, IL-6, IL-1β, macrophage inflammatory protein (MIP)-1α, MIP-1β, monocyte chemotactic protein-1, intercellular adhesion molecule-1, surfactant protein (SP)-D, granulocyte macrophage colony-stimulating factor, IL-23, IL-33, IL-25, IL-10, albumin, and protein
Exhaled particles IL-6 and IL-8 | Day 21 (±2 days)
Blood inflammatory markers including C-reactive protein, TNF-α, IL-6, IL-8, and α2-macroglobulin | Day 21 (±2 days)
Plasma EP395 | Day 7 (±2 days) [only applicable for trough levels of EP395], Day 14 (±2 days) and Day 21 (±2 days)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hohlfeld, Prof. Dr., Principal Investigator — Fraunhofer Institute for Toxicology and Experimental Medicine ITEM
Locations (1):
- Fraunhofer Institute for Toxicology and Experimental Medicine ITEM, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No